CLINICAL TRIAL: NCT06484491
Title: Radiotherapy Dose Escalation Using Intensity-modulated Proton Therapy for Non-small-cell Lung Cancer Patients
Brief Title: IMPT Dose Escalation for NSCLC (HyDose)
Acronym: HyDose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNM16745; NL86435.042.24 (Other: CCMO register)
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Neoplasms; Proton Therapy; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Carboplatin; Pemetrexed; Induction Chemotherapy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 Intervention group (Experimental): Dose-escalated IMPT
  Interventions: Radiation: Dose-escalated intensity-modulated proton therapy (IMPT-74); Drug: Cisplatin or carboplatin + pemetrexed for induction chemotherapy, cisplatin + docetaxel for concurrent chemotherapy; Drug: Immunotherapy: adjuvant durvalumab

INTERVENTIONS:
Radiation: Dose-escalated intensity-modulated proton therapy (IMPT-74) — Heterogeneous simultaneous integrated boost of 74.0 Gy (RBE) to primary tumor >15mm away form mediastinal envelope, and 64.0 Gy (RBE) to primary tumor =< 15mm away from mediastinal envelope. The rest of the clinical target volume, including affected lymph nodes, receives 60.0 Gy (RBE).
Drug: Cisplatin or carboplatin + pemetrexed for induction chemotherapy, cisplatin + docetaxel for concurrent chemotherapy — Induction course:
  -Cisplatin (75 mg/m2) or carboplatin (AUC 6) + pemetrexed (500mg/m2).
  Concurrent chemoradiotherapy:
  * Weekly cisplatin (20mg/m2) + docetaxel (20mg/m2) on Mondays.
  * Radiotherapy will be given for 5x5 days.
Drug: Immunotherapy: adjuvant durvalumab — Adjuvant treatment will be given starting 1-6 weeks after chemoradiotherapy if no progression, good performance (PS 0-1), no other contra-indication for immunotherapy.
  Doses:
  * Start durvalumab 10 mg/kg 1x/14 days.
  * If possible after 2 courses switch to 1500 mg flat dose 1x/4 wk.
  * Continue for 12 months in total.

SUMMARY:
The goal of this clinical pilot trial is to learn if dose to the tumor in the lung can be safely increased using proton therapy in stage III non-small-cell lung cancer patients receiving combined chemotherapy and radiotherapy. The main questions it aims to answer are:

* Is the risk of severe radiotherapy toxicities (requiring hospital admission) within acceptable margins ?
* What is a rough estimate of the effect of the treatment under study?

Compared to standard care in our clinic, all participants in this pilot trial will

* Receive a higher dose of proton therapy to the tumor in the lung albeit with the same number of radiotherapy visits as the current standard treatment.
* Receive two additional follow-up visits at the clinic after treatment, namely 4 and 6 weeks after finishing radiotherapy.
* Two additional blood withdrawals at the last week of radiotherapy and 4 weeks after finishing radiotherapy, to measure a type of white blood cells.
* Receive an extra quality of life questionnaire at the last week of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* WHO performance score 0-2
* Histologically proven stage III NSCLC
* Planned for CCRT and adjuvant immunotherapy (intention to treat)
* Primary tumour volume outside of mediastinal PRV (i.e., mediastinal envelope + 5 mm) ≥60% of total primary tumour volume (true for 75% of patients in preliminary analysis), for sufficient dose escalation

Exclusion Criteria:

* Chemotherapy not given concurrently with radiotherapy
* Upfront decision that adjuvant immunotherapy is not possible
* Primary tumour overlapping ≥40% with mediastinal PRV
* Unable or unwilling to understand the information on trial-related topics, to give informed consent or to fill out quality-of-life questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Severe (grade 3+) adverse effects up to six months after radiotherapy | Data for assesing safety will be recorded from day 1 to 365

SECONDARY OUTCOMES:
Local control of the lung tumour assessed by the treating physician and radiologist according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Data for assessing local control will be recorded up to 2 years after chemoradiotherapy
  Local control was defined as the time from randomization until the date of objective disease progression in the lungs (RECIST 1.1). Local progression was defined using RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Local control was calculated using the Kaplan-Meier technique.
Progression-free survival based on review by the treating physician and radiologist according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Data for assessing progression-free survival will be recorded up to 2 years after chemoradiotherapy
  PFS was defined as the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression). Progression was defined using RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PFS was calculated using the Kaplan-Meier technique.
Distant metastasis control based on review by the treating physician and radiologist according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Data for assessing distant metastasis will be recorded up to 2 years after chemoradiotherapy
  Time to distant metastasis was defined as the time from the date of randomization until the first date of distant metastasis. Distant metastasis was defined as any new lesion that was outside of the radiation field according to RECIST 1.1 or proven by biopsy. Time to distant metastasis was calculated using the Kaplan-Meier technique.
Overall survival | Data for assessing overall survival will be recorded up to 2 years after chemoradiotherapy
Grade 2+ adverse effects (i.e., requiring medication), both acute and late | Data for assesing safety will be recorded from day 1 to 365
Qualifying for adjuvant immunotherapy after finishing chemoradiotherapy yes/no | Data on qualifying for adjuvant immunotherapy will be recorded up to 6 weeks after finishing chemoradiotherapy
European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30) | Data for assesing quality of life will be recorded up to day 730
  The EORTC QLQ-C30 is a disease specific measurement instrument for use in patients with or cured from cancer. It measures a number of aspects of quality of life, namely: physical functioning; role functioning; emotional functioning; cognitive functioning; social functioning. It also evaluates symptoms, such as pain, nausea, sleep, dyspnea, cancer related fatigue, and constipation, diahorrea, and fincancial problems, as well as two questionas about overall quality of life.
  The questionnaire consists of a total of 30 items, divided over 9 subscales. The items are on Likert scales. The scores for each subscale can be calculated on a 0-100 scale, as well as the total score. A high score for a functional scale represents a high/healthy level of functioning. A high score for global health status / QoL represents a high QoL. By contrast, a high score for a symptom scale/item represents a high level of symptomatology/problems.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Lung Cancer 13-item (EORTC-QLQ-LC13) | Data for assesing quality of life will be recorded up to day 730
  The EORTC QLQ-LC13 is a 13-item lung cancer-specific questionnaire module meant as a disease-specific extension to the EORTC QLC-C30. It contains both multi-item (dyspnea) and single-item (all others) measures of lung cancer-associated symptoms (i.e. coughing, haemoptysis, dyspea and pain) and side-effects from conventional chemo- and radiotherapy (i.e. hair loss, neuropathy, sore mouth and dysphagia). The items are scored on likert scales, and can be converted to a 0-100 scale for each symptom and side effect. A high score represents a high level of symptomatology or problems.
3 EuroQoL-5D three-level version (EQ-5D-3L) | Data for assesing quality of life will be recorded up to day 730
  This questionnaire consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale (EQ VAS):
  * The descriptive system comprises five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems, extreme problems (labelled 1-3). The respondent indicates their health by checking the box against the most appropriate statement in each of the five dimensions.
  * The EQ VAS redords the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Lymphocyte counts after finishing chemoradiotherapy | Data for assessing lymphocyte counts will be assessed between 4 and 6 weeks after chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: R. Wijsman, MD PhD, Principal Investigator — University Medical Center Groningen; A. Van der Wekken, MD PhD, Principal Investigator — University Medical Center Groningen; E. Korevaar, dr ir (PhD), Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands